CLINICAL TRIAL: NCT00003110
Title: A Phase II Trial of 72-Hour Continuous Infusion Bleomycin as Salvage Therapy in AIDS-Related and Immunocompetent Non-Hodgkin's Lymphoma
Brief Title: Bleomycin in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Scot C. Remick, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU5496; P30CA043703 (NIH); CWRU-5496 (Other: Case Comprehensive Cancer Center); AMC-7A-94; BMS-CWRU-5496; NCI-G97-1343
Record Dates: First submitted 1999-11-01; First posted 2004-04-07 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Lymphoma
Keywords: recurrent childhood lymphoblastic lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related diffuse large cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related small noncleaved cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell | interventions — Bleomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: bleomycin sulfate — Patients receive bleomycin by continuous infusion for 72 hours every 3 weeks. Induction therapy consists of 3 cycles. Patients who achieve complete remission receive 2 more cycles. Patients with partial remission or stable disease may continue therapy until disease progression or unacceptable toxicity occurs.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of bleomycin in treating patients with non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate, response duration and survival of patients receiving bleomycin as salvage therapy for AIDS-related or immunocompetent non-Hodgkin's lymphoma. II. Assess the feasibility and toxicity of treatment for this disease. III. Evaluate the quality of life of AIDS and non-AIDS patients with non-Hodgkin's lymphoma.

OUTLINE: Patients are stratified by number of prior cytotoxic chemotherapy regimens, prior radiotherapy, and HIV/AIDS status. Patients receive bleomycin by continuous infusion for 72 hours every 3 weeks. Induction therapy consists of 3 cycles. Patients who achieve complete remission receive 2 more cycles. Patients with partial remission or stable disease may continue therapy until disease progression or unacceptable toxicity occurs. Quality of life assessments are conducted at beginning of therapy, every 3 weeks, and at completion of treatment. Patients are followed every 3 months for overall survival.

PROJECTED ACCRUAL: A total of 32 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent intermediate or high grade non-Hodgkin's lymphoma (NHL) AIDS-related NHL eligible At least 1 evaluable or measurable disease as defined by the following: Radiographic findings are acceptable Bidimensionally measurable defect on a computed tomographic (CT) scan Clearly defined abdominal masses on CT scans Enlarged spleen and/or liver extending at least 5 cm below the costal margin Biopsy proven lymphomatous hepatic involvement No clinical or radiographic evidence of parenchymal CNS involvement by lymphoma (meningeal lymphoma permitted) A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: Any age Performance status: ECOG 0-3 Life expectancy: At least 6 weeks Hematopoietic: WBC at least 1500/mm3 Platelet count at least 50,000/mm3 Hepatic: Bilirubin no greater than 3.0 mg/dL Renal: Creatinine no greater than 3.0 mg/dL Other: May be HIV positive Immunocompetent (HIV-seronegative) NHL patients must be suitable candidates for bleomycin chemotherapy Active infections undergoing drug treatment allowed Negative head CT/MRI scan

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 1 prior systemic chemotherapy regimen Endocrine therapy: Not specified Radiotherapy: Prior radiation therapy for localized stage I/II disease that has progressed beyond initial radiation therapy port is allowed Surgery: Not specified Other: Concurrent zidovudine, didanosine, or zalcitabine therapy allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1997-07; Primary Completion 2001-08 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
The effectiveness of bleomycin in treating patients with non-Hodgkin's lymphoma. | Continuous infusion for 72 hours every 3 weeks. Induction therapy consists of 3 cycles. Patients who achieve CR receive 2 more cycles. Patients with PR or stable disease may continue therapy until disease progression or unacceptable toxicity occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Scot C. Remick, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States